CLINICAL TRIAL: NCT03912324
Title: Computed Tomogram Myocardial Thickness Map Guided pulmOnary Vein iSolaTion vs. Empirical Pulmonary Vein Isolation in Cryoballoon Ablation for Paroxysmal Atrial Fibrillation (UTMOST AF II)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0109
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial fibrillation; Pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unipolar voltage subtraction map guided PV isolation group (Experimental): 1. Pulmonary vein isolation will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury
  3. Mapping of echocardiographic unipolar voltage subtraction after atrial septal puncture
  4. the electrode map data is transferred to the core lab by network to calculate the unipolar voltage subtraction color map (within 10 minutes)
  5. Increase radiofrequency ablation time by 2 to 5 seconds in areas with high potential in unipolar voltage subtraction color map
  6. Decrease radiofrequency ablation time by 2 to 5 seconds in areas with low potential in unipolar voltage subtraction color map
  7. Evaluation of success rate and time of pulmonary vein isolation after bilateral pulmonary vein primary columnar resection
  8. Evaluate time to complete isolation after additional ablation
  9. Evaluation of Procedure and Ablation time, and perfusion saline dose
  10. Rhythm follow-up after the procedure in accordance with the study design.
  Interventions: Procedure: Unipolar voltage subtraction map guided PV isolation group
- CT myocardial thickness map guided PV isolation group (Experimental): 1. Pulmonary vein isolation will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. Prepared myocardial thickness map with CT DICOM images conducted prior to procedure.
  4. Increase radiofrequency ablation time by 2 to 5 seconds in thick areas in CT myocardial thickness map
  5. Decrease radiofrequency ablation time by 2 to 5 seconds in thin areas in CT myocardial thickness map
  6. Evaluation of success rate and time of pulmonary vein isolation after bilateral pulmonary vein primary columnar resection
  7. Evaluate time to complete isolation after additional ablation
  8. Evaluation of Procedure time, Ablation time, and perfusion saline dose
  9. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Interventions: Procedure: CT myocardial thickness map guided PV isolation group
- Empirical PV isolation group (Active Comparator): 1. Pulmonary vein isolation will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. The procedure is performed by adjusting radiofrequency energy according to the traditional method and experience of the practitioner.
  4. Evaluation of success rate and time of pulmonary vein isolation after bilateral pulmonary vein primary columnar resection
  5. Evaluate time to complete isolation after additional ablation
  6. Evaluation of Procedure time, Ablation time, and perfusion saline dose
  7. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Interventions: Procedure: Empirical PV isolation group

INTERVENTIONS:
Procedure: Unipolar voltage subtraction map guided PV isolation group — 1. Pulmonary vein isolation will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury
  3. Mapping of echocardiographic unipolar voltage subtraction after atrial septal puncture
  4. the electrode map data is transferred to the core lab by network to calculate the unipolar voltage subtraction color map (within 10 minutes)
  5. Increase radiofrequency ablation time by 2 to 5 seconds in areas with high potential in unipolar voltage subtraction color map
  6. Decrease radiofrequency ablation time by 2 to 5 seconds in areas with low potential in unipolar voltage subtraction color map
  7. Evaluation of success rate and time of pulmonary vein isolation after bilateral pulmonary vein primary columnar resection
  8. Evaluate time to complete isolation after additional ablation
  9. Evaluation of Procedure and Ablation time, and perfusion saline dose
  10. Rhythm follow-up after the procedure in accordance with the study design.
  Arms: Unipolar voltage subtraction map guided PV isolation group
Procedure: CT myocardial thickness map guided PV isolation group — 1. Pulmonary vein isolation will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. Prepared myocardial thickness map with CT DICOM images conducted prior to procedure.
  4. Increase radiofrequency ablation time by 2 to 5 seconds in thick areas in CT myocardial thickness map
  5. Decrease radiofrequency ablation time by 2 to 5 seconds in thin areas in CT myocardial thickness map
  6. Evaluation of success rate and time of pulmonary vein isolation after bilateral pulmonary vein primary columnar resection
  7. Evaluate time to complete isolation after additional ablation
  8. Evaluation of Procedure time, Ablation time, and perfusion saline dose
  9. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: CT myocardial thickness map guided PV isolation group
Procedure: Empirical PV isolation group — 1. Pulmonary vein isolation will be performed using a radiofrequency catheter
  2. Esophageal temperature will be monitored to prevent esophageal injury.
  3. The procedure is performed by adjusting radiofrequency energy according to the traditional method and experience of the practitioner.
  4. Evaluation of success rate and time of pulmonary vein isolation after bilateral pulmonary vein primary columnar resection
  5. Evaluate time to complete isolation after additional ablation
  6. Evaluation of Procedure time, Ablation time, and perfusion saline dose
  7. Rhythm follow-up will be performed after the procedure in accordance with the aforementioned study design.
  Arms: Empirical PV isolation group

SUMMARY:
New parameters or methods, such as ablation index, have been developed for the quantification of high-frequency energy used in pulmonary vein isolation, but there is no known method for atrial fibrillation considering individual differences in atrial tissue. The atrium is only 1/3 of the thickness of the ventricle and is thinner in women and older than men or young people.

The aim of this study was to evaluate the efficacy and safety of radiofrequency energy therapy using atrial individual differences. In order to reflect the thickness of the atrium, we will use the unipolar and bipolar maps and the myocardial thickness map using computed tomography (CT) images. To evaluate the efficacy and safety of energy titration therapy by random assignment of high frequency energy therapy group, CT image application high frequency energy therapy group, and existing empirical high frequency therapy group.

DETAILED DESCRIPTION:
A. Study design

1. Prospective randomization (Unipolar voltage subtraction map guided PV(pulmonary vein) isolation group vs. CT myocardial thickness map guided PV isolation group vs. Empirical PV isolation group )
2. Target number of subjects: 480 (160 per group)
3. Rhythm FU : 2012 ACC/AHA/ESC guidelines (Holter monitoring at the baseline, 2 month, and thereafter every 6 months; ECG if the patient has any symptom)
4. Anticoagulant therapy followed by 2014 ACC/AHA/ESC guidelines
5. All complications in each group will be evaluated including the re-hospitalization rate, major cardiovascular event, and mortality rate.

B. Progress and rhythm/ECG follow-up

1. To be performed in accordance with the 2012 ACC/AHA/HRS guidelines for AF management
2. Follow-up at 1 weeks, 3 months, and thereafter every 6-month after procedure.
3. Rhythm control at 3 months, and thereafter every 6-month follow-up with Holter
4. If the patient complains of symptoms, ECG will be performed at any time, and rhythm follow-up will be carried out with a Holter or event recorder.

C. Follow-up All the patients will be followed-up at 1, 3, 6 months, and thereafter every 6 months. If the patient shows any symptom within the clinical study period, patient will visit the outpatient clinic. ECG will be performed at every outpatient visits, and 24-hour Holter or event recording will be performed every 6 months for 2 years, and every year after 2 years (2012 Heart Rhythm Society/EHRA/European Cardiac Arrhythmia Society Expert Consensus Statement guidelines). If atrial fibrillation or atrial tachycardia lasting more than 30 seconds is observed in 12-lead ECG or Holter, it will be evaluated as recurrence. Recurrence within 3 months after the procedure will be classified as early recurrence, and that after 3 months will be classified as clinical recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with paroxysmal atrial fibrillation who is scheduled for ablation procedure and ≥20 and ≤80 years of age
2. Left atrium size < 50mm
3. paroxysmal atrial fibrillation that is recurrence during antiarrhythmic drug treatment or is not able to use an antiarrhythmic drug.
4. Patient who is indicated for anticoagulation therapy (for prevention of cerebral infarction)

Exclusion Criteria:

1. Patients with persistent or permanent atrial fibrillation
2. Atrial fibrillation associated with severe cardiac malformation or a structural heart disease that is hemodynamically affected
3. Patients with severe renal impairment or CT imaging difficulty using contrast media
4. Patients with a past history of radiofrequency ablation for atrial fibrillation or other cardiac surgery
5. Patients with active internal bleeding
6. Patients with contraindications for anticoagulation therapy(for prevention of cerebral infarction) and antiarrhythmic drugs
7. Patients with valvular atrial fibrillation (mitral stenosis >grade 2, mechanical valve, mitral valvuloplasty)
8. Patients with a severe comorbid disease
9. Expected survival < 1 year
10. Drug addicts or alcoholics
11. Patients who cannot read the consent form (illiterates, foreigners, etc.)
12. Other patients who are judged by the principal or sub-investigator to be ineligible for participation in this clinical study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation: Procedure-related cardiac complication rate | within 30 days post procedure
  including open cardiac surgery, cerebral infarction, pericardial effusion or cardiac tamponade, hematoma in the inguinal puncture site and vascular complications within 30 days post procedure.
Efficacy evaluation: Atrial fibrillation or atrial tachycardia for at least 30 seconds after 3 months within 1 year without antiarrhythmic medication | Within 1 year after 3 months of procedure
  Defined as atrial fibrillation or atrial tachycardia > 30 sec after 3 months within 1 year; based on the 2012 ACC/AHA/HRS guidelines, 24-hour Holter ECG monitoring will be performed at 2 month and every 6 months, and ECG and monitoring with a Holter or an event recorder will be performed at any time if the patient complains of symptoms
Efficacy evaluation: Major cardiovascular event rate | immediate after procedure
  death, myocardial infarction, coronary angioplasty, and re-hospitalization for arrhythmia and heart failure
Efficacy evaluation: Major cardiovascular event rate | 12 months after procedure
  death, myocardial infarction, coronary angioplasty, and re-hospitalization for arrhythmia and heart failure

SECONDARY OUTCOMES:
Comparison of procedure time | immediate after procedure
Comparison of ablation time | immediate after procedure
Comparison of hospitalization period | immediate after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 1 week after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 3 months after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 6 months after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 12 months after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 18 months after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 24 months after procedure
Comparison of anti-arrhythmic drug or anticoagulation therapy related complication rate | 36 months after procedure
Comparison of re-hospitalization rate after the procedure | 1 week after procedure
Comparison of re-hospitalization rate after the procedure | 3 months after procedure
Comparison of re-hospitalization rate after the procedure | 6 months after procedure
Comparison of re-hospitalization rate after the procedure | 12 months after procedure
Comparison of re-hospitalization rate and number of electrical cardioversion after the procedure | 18 months after procedure
Comparison of re-hospitalization rate after the procedure | 24 months after procedure
Comparison of re-hospitalization rate after the procedure | 36 months after procedure
Comparison of number of electrical cardioversion after the procedure | 1 week months after procedure
Comparison of number of electrical cardioversion after the procedure | 3 months after procedure
Comparison of number of electrical cardioversion after the procedure | 6 after procedure
Comparison of number of electrical cardioversion after the procedure | 12 months after procedure
Comparison of number of electrical cardioversion after the procedure | 18 months after procedure
Comparison of number of electrical cardioversion after the procedure | 24 months after procedure
Comparison of number of electrical cardioversion after the procedure | 36 months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No